CLINICAL TRIAL: NCT01743807
Title: A Phase I Study of GNKG168 in Pediatric Patients With Acute Lymphoblastic Leukemia or Acute Myeloid Leukemia (IND#113600)
Brief Title: Phase I Study of GNKG168 in Acute Lymphoblastic Leukemia and Acute Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: SBI Biotech (supplier) decided to no longer support the study or GNKG168.
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: SBI Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Nobuko Hijiya, MD, Associate Professor of Pediatrics, Therapeutic Advances in Childhood Leukemia Consortium
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2009-008
Record Dates: First submitted 2012-11-28; First posted 2012-12-06 (Estimated); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Relapsed Acute Lymphoblastic Leukemia; Relapsed Acute Myelogenous Leukemia
Keywords: Relapsed; Minimal Residual Disease; MRD; Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; ALL; AML; GNKG168; Pediatric; Childhood
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Recurrence; Neoplasm, Residual | interventions — GNKG168

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Post-HSCT (Experimental): Patients who have a history of hematopoetic stem cell transplantation (HSCT). GNKG168 will be administered as a 60 minute intravenous infusion daily for 5 consecutive days. It may be repeated every 14 days. Patients should receive minimum 2 courses and up to 6 courses may be administered. Dose will be assigned at study entry.
  Interventions: Drug: GNKG168
- No HSCT (Experimental): Patients who have never undergone HSCT. GNKG168 will be administered as a 60 minute intravenous infusion daily for 5 consecutive days. It may be repeated every 14 days. Patients should receive minimum 2 courses and up to 6 courses may be administered. Dose will be assigned at study entry.
  Interventions: Drug: GNKG168

INTERVENTIONS:
Drug: GNKG168 — GNKG168 will be given intravenously over 1 hour on days 1 through 5 followed by 9 days of rest. Dose will be assigned at study entry.
  Dose Level 0: 0.15 mg/kg Dose Level 1: 0.25 mg/kg Dose Level 2: 0.75 mg/kg Dose Level 3: 1.5 mg/kg
  The starting dose level for the trial will be 0.25 mg/kg. If that dose level proves to be intolerable, the dose will be reduced to 0.15 mg/kg (dose level 0). If the 0.15 mg/kg dose level is intolerable due to DLTs, TACL, the Principal Investigator, and Medical Monitor will then decide the best course of action for subsequent administration of GNKG168.
  Other Names: CpG685

SUMMARY:
This is a phase I trial of an investigational drug called GNKG168 in patients with relapsed and refractory acute lymphoblastic leukemia (ALL) and acute myelogenous leukemia (AML) who are in morphologic remission but are positive for Minimum Residual Disease (MRD).

DETAILED DESCRIPTION:
GNKG168 is a Toll-like receptor (TLR) agonist. TLR agonists are a novel approach to stimulate an effective anti-tumor immune response as they are able to stimulate both innate and adaptive immune responses. There will be two strata i.e patients who have received hematopoietic stem cell transplant (HSCT) and patients who have never undergone HSCT. GNKG168 will be administered as a 60 min iv infusion. One 14-day cycle consists of 5-day treatment followed by 9 day-rest. Patients will receive 2 cycles before evaluation. The primary objective is to determine the maximum tolerated dose of GNKG168 in relapsed ALL and AML patients. The completion of this study and the correlative studies will provide a solid foundation for subsequent phase 2 study and the development of clinical applications of CpG-ODN-based immune therapy as a treatment of childhood leukemia. If safety and efficacy of GNKG168 is proven, it will be intriguing to explore its role to maintain CR in a randomized manner.

ELIGIBILITY:
Inclusion Criteria

1. Age Patients must be ≥1 and ≤ 21 years of age when originally diagnosed with ALL or AML.
2. Diagnosis

   1. Patients must have previously histologically confirmed ALL or AML at original diagnosis or previous relapse. Patients with treatment-related AML are eligible.
   2. Patients must be in complete remission (CR) with less than 5% blasts in the bone marrow.

      * Post-HSCT patients should be in first or greater CR
      * Patients who have never received HSCT should be in second or greater CR
   3. Patient must have detectable MRD (≥0.01%) by flow cytometry.
3. Performance Level Karnofsky ≥ 50% for patients >16 years of age and Lansky ≥ 50% for patients ≤16 years of age.
4. Prior Therapy

   1. Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy.
   2. At least 14 days must have elapsed since any treatment with systemic chemotherapy including high-dose steroid (prednisone>0.5 mg/kg or equivalent), radiotherapy, biological therapy or any other investigational therapy. (Note: low-dose steroid; prednisone ≤0.5 mg/kg/day or equivalent is allowed.)
   3. At least 28 days must have elapsed since any cellular therapies such as chimeric antigen receptor-modified T cells.
   4. Patients who have never had HSCT must not be a suitable candidate for HSCT. For this protocol, a suitable candidate is defined as one who has an identified donor with plans to undergo transplant within the next 28 days.
   5. Previous HSCT:

      * Patients having received HSCT are eligible and 60 days must have elapsed since stem cell infusion.
      * Patients having received donor lymphocyte infusions (DLI) are eligible.
      * At least 28 days must have elapsed from the last DLI.
      * Must have ≥90% donor chimerism. The test for donor chimerism must have been done within the last 60 days. If patient has subsequently relapsed after HSCT but prior to enrollment on this study, the donor chimerism test is not needed.
      * Patients must have been off all immune suppression drugs for 7 days before study entry. (at least 2 weeks for high-dose steroid, i.e. prednisone>0.5 mg/kg or equivalent; see 4b above) (Note; low-dose steroid; prednisone ≤0.5 mg/kg/day or equivalent is allowed.)
5. Renal and Hepatic Function

   1. Patients must have a serum creatinine that is less than or equal to 1.5 x the institutional upper limit of normal according to age. (Grade 1 per the CTCAE 4.0)
   2. Patient's ALT and AST must be less than or equal to 3 x institutional upper limit of normal. (Grade 1 per the CTCAE 4.0)
   3. Patient's total bilirubin must be less than or equal to 1.5 x institutional upper limit of normal. (Grade 1 per the CTCAE 4.0)
6. Cardiac Function Patient must have a shortening fraction > 27% by ECHO or an ejection fraction > 45% by MUGA.
7. Reproductive Function

   1. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
   2. Female patients with infants must agree not to breastfeed their infants while on this study.
   3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.
8. Hematological Function Patients must have an absolute neutrophil count > 750/dL, platelets > 75,000/dL AND absolute lymphocyte count > 200/uL which is not decreasing. Patients with previous HSCT may have a platelet count > 50,000/dL.

Exclusion Criteria

Patients will be excluded if they meet any of the following criteria.

1. Graft versus host disease (GVHD) that meets the following criteria:

   1. Active grade 2 or higher acute GVHD at the time of study entry.
   2. Active chronic GVHD (moderate or severe).
2. Plan for donor lymphocyte infusions during the study period.
3. Need for immunosuppressive medications including high-dose corticosteroids (prednisone >0.5 mg/kg or equivalent) (Note: low-dose steroid; prednisone ≤0.5 mg/kg/day or equivalent is allowed.)
4. Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
5. Patient will be excluded if they are currently receiving other investigational drugs.
6. Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
7. Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with the prescribed protocol therapy, interfere with consent, study participation, follow up, or interpretation of study results.
8. Patients with CNS 3 disease are excluded. No CNS therapy will be allowed during the first 2 courses of therapy.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2014-07-28 (Actual); Study Completion 2014-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuko Hijiya, MD, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago; Kirk Schultz, MD, Study Chair — British Columbia Children's Hospital
Locations (3):
- United States (3):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Groups:
- Post HSCT- Dose Level 0; Post HSCT- Dose Level 1; Post HSCT- Dose Level 2; Post HSCT- Dose Level 3: Hematopoietic stem cell transplantation (HSCT)
  Dose level 0: 0.15 mg/kg/dose Dose level 1: 0.25 mg/kg/dose Dose level 2: 0.75 mg/kg/dose Dose level 3: 1.5 mg/kg/dose
- No HSCT- Dose Level 0; No HSCT- Dose Level 1; No HSCT- Dose Level 2; No HSCT- Dose Level 3: No HSCT: Never had a Hematopoietic stem cell transplantation (HSCT)
  Dose level 0: 0.15 mg/kg/dose Dose level 1: 0.25 mg/kg/dose Dose level 2: 0.75 mg/kg/dose Dose level 3: 1.5 mg/kg/dose
Period: Overall Study
Arm/Group | Post HSCT- Dose Level 0 | Post HSCT- Dose Level 1 | Post HSCT- Dose Level 2 | Post HSCT- Dose Level 3 | No HSCT- Dose Level 0 | No HSCT- Dose Level 1 | No HSCT- Dose Level 2 | No HSCT- Dose Level 3
Started | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Completed ("Completed" is defined here as completing 1 or more courses of therapy.) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The total number of enrolled subjects were 3. One HSCT patient enrolled on dose level #1, and two non-HSCT patients enrolled onto dose level #1.
Groups:
- HSCT Dose Level 0: Hematopoietic stem cell transplantation (HSCT)
  Dose level 0: 0.15 mg/kg/dose Dose level 1: 0.25 mg/kg/dose Dose level 2: 0.75 mg/kg/dose Dose level 3: 1.5 mg/kg/dose
- HSCT Dose Level 1; HSCT Dose Level 2; HSCT Dose Level 3: Hematopoietic stem cell transplantation (HSCT)
- Non-HSCT Dose Level 0: No HSCT: Never had a Hematopoietic stem cell transplantation (HSCT)
  Dose level 0: 0.15 mg/kg/dose Dose level 1: 0.25 mg/kg/dose Dose level 2: 0.75 mg/kg/dose Dose level 3: 1.5 mg/kg/dose
- Non-HSCT Dose Level 1; Non-HSCT Dose Level 2; Non-HSCT Dose Level 3: No HSCT: Never had a Hematopoietic stem cell transplantation (HSCT)
- Total: Total of all reporting groups
Arm/Group | HSCT Dose Level 0 | HSCT Dose Level 1 | HSCT Dose Level 2 | HSCT Dose Level 3 | Non-HSCT Dose Level 0 | Non-HSCT Dose Level 1 | Non-HSCT Dose Level 2 | Non-HSCT Dose Level 3 | Total
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Between 18 and 65 years | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Male | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Prior Hematopoetic Stem Cell Transplantation (HSCT) [Count of Participants; unit: Participants] | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT) in the First Two Courses of Therapy
Description: DLT is defined as:
  A) Any non-hematologic toxicity that is ≥ CTCAE grade 3 and at least possibly related to GNKG168 (the relationship to GNKG168 cannot be ruled out), with the EXCEPTION of the following toxicities when observed at Grade 3:
  * Fatigue
  * Fever
  * Anorexia
  * Rash that turns to grade ≤ 2 within 7 days
  * Elevation in hepatic transaminases (ALT/SGOT and AST/SGPT), GGT or alkaline phosphatase that returns to ≤ grade 2 within 14 days. It will not be considered a DLT if the patient exits the study and begins alternative therapy before the end of the 14 day evaluation period.
  B) Grade 3 or 4 hematologic toxicity that is at least possibly related to GNKG168 that does not reverse to baseline within 7 days.
  C) For patients who have undergone HSCT, DLT will include the onset of Grade 3 or 4 acute GVHD, the onset of moderate to severe chronic GVHD, the onset of bronchiolitis obliterans and graft failure.
Time Frame: Beginning with the first dose of GNKG168 until the end of course 2; courses are 14 days so there will be approximately 28 days of monitoring for DLT
Population: Immunomodulatory molecules were examined at two time points. Analyses were limited to the pretreatment and first post treatment samples. Additional samples were excluded from the analysis. A paired t-test was performed to examine the effect of first treatment on the expression of each gene in the CodeSet. Significance was declared at a nominal p-value threshold of 0.05. We note that this liberal p-value threshold was chosen due to the limited sample size.
Measure: Count of Participants; unit: Participants
Groups:
- Post HSCT- Dose Level 1: Hematopoietic stem cell transplantation (HSCT)
  Dose level 1: 0.25 mg/kg/dose
- Post HSCT- Dose Level 2: Hematopoietic stem cell transplantation (HSCT)
  Dose level 2: 0.75 mg/kg/dose
- Post HSCT- Dose Level 3: Hematopoietic stem cell transplantation (HSCT)
  Dose level 3: 1.5 mg/kg/dose
- No HSCT- Dose Level 1: No HSCT: Never had a Hematopoietic stem cell transplantation (HSCT)
  Dose level 1: 0.25 mg/kg/dose
- No HSCT- Dose Level 2: No HSCT: Never had a Hematopoietic stem cell transplantation (HSCT)
  Dose level 2: 0.75 mg/kg/dose
- No HSCT- Dose Level 3: No HSCT: Never had a Hematopoietic stem cell transplantation (HSCT)
  Dose level 3: 1.5 mg/kg/dose
Arm/Group | Post HSCT- Dose Level 0 | Post HSCT- Dose Level 1 | Post HSCT- Dose Level 2 | Post HSCT- Dose Level 3 | No HSCT- Dose Level 0 | No HSCT- Dose Level 1 | No HSCT- Dose Level 2 | No HSCT- Dose Level 3
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Post HSCT- Dose Level 2 vs No HSCT- Dose Level 1 vs No HSCT- Dose Level 3; Test type: Superiority; p = 0.05, t-test, 2 sided

2. Secondary Outcome: The Number of Participants With a Decrease in Minimal Residual Disease (MRD) Present in Patients Treated With GNKG168
Description: Doctors have developed a test to detect very small amounts of leukemia that still exist even though it looks like remission under a microscope. This test is called Minimal Residual Disease (MRD). MRD is very specific and can detect 1 cancer cell out of 10,000 regular cells. The results of the MRD test on bone marrow can show when a patient has a very small amount of cancer cells left in the bone marrow. We will use this test to evaluate the effect of GNKG168 in killing the small amount of cells left in your bone marrow.
Time Frame: Pre-study and End of Course 1 (Day 14)
Population: Patients who had MRD analyzed at both the pre-study event and end of course 1.
Measure: Count of Participants; unit: Participants
Groups:
- HSCT- Dose Level 0: Hematopoietic stem cell transplantation (HSCT)
  Dose level 0: 0.15 mg/kg/dose Dose level 1: 0.25 mg/kg/dose Dose level 2: 0.75 mg/kg/dose Dose level 3: 1.5 mg/kg/dose
- HSCT- Dose Level 1: Hematopoietic stem cell transplantation (HSCT)
  Dose level 1: 0.25 mg/kg/dose
- HSCT- Dose Level 2: Hematopoietic stem cell transplantation (HSCT)
  Dose level 2: 0.75 mg/kg/dose
- HSCT- Dose Level 3: Hematopoietic stem cell transplantation (HSCT)
  Dose level 3: 1.5 mg/kg/dose
Arm/Group | HSCT- Dose Level 0 | HSCT- Dose Level 1 | HSCT- Dose Level 2 | HSCT- Dose Level 3 | No HSCT- Dose Level 0 | No HSCT- Dose Level 1 | No HSCT- Dose Level 2 | No HSCT- Dose Level 3
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Occurrence of Graft Versus Host Disease (GVHD) in Patients Who Had Previous HSCT and Received GNKG168
Description: We will evaluate the impact of GNKG168 on induction of clinical GVHD using the consensus scoring system developed by NIH (Filipovich et. al., National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. Diagnosis and Staging Working Group Report, Biology of Blood and Marrow Transplantation, Volume 11, Issue 12, Dec. 2005, pp. 945-956)
Time Frame: Weekly during Courses 1 and 2 (i.e, 4 times in 28 days), Day 1 of Courses 3-6 (approximately Days 29, 43 and 57), and when patient is removed from protocol therapy.
Population: 2 HSCT patients enrolled in dose level #1,one of the patients never began treatment as was no longer eligible for treatment due to peripheral blasts. Therefore 1 patient was enrolled and completed treatment at dose level 1. There were 2 Non-HSCT patients enrolled at dose level 1 who completed the treatment.
Measure: Count of Participants; unit: Participants
Groups:
- HSCT- Dos level1: Hematopoietic stem cell transplantation (HSCT)
  Dose level 1: 0.25 mg/kg/dose
Arm/Group | HSCT- Dose Level 0 | HSCT- Dos level1 | HSCT- Dose Level 2 | HSCT- Dose Level 3 | No HSCT- Dose Level 0 | No HSCT- Dose Level 1 | No HSCT- Dose Level 2 | No HSCT- Dose Level 3
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Occurrence of Graft Failure in Patients Who Previously Had a HSCT and Received GNKG168
Description: Peripheral blood samples will be evaluated for the presence of cGVHD biomarkers. Change in level of MRD, and MRD response following GNKG168
Time Frame: Day 14
Population: Study terminated early and the variable was not analyzed.
Groups:
- HSCT Participants Who Received Treatment: Participants with prior HSCT who received protocol therapy
Arm/Group | HSCT Participants Who Received Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in the Percent of ALL or AML Blasts Exhibiting Markers of Immunogenicity and Apoptosis
Description: Change in the percent of ALL or AML blasts exhibiting markers of immunogenicity and apoptosis will be analyzed from bone marrow specimens.
Time Frame: End of Course 1 (Day 14), end of Course 2 (approx. Day 28), end of courses 4 and 6 (approx. Days 56 and 70), and date removed from therapy if previous marrow sample > 2 weeks ago
Population: Study terminated early and the variable was not analyzed.
Groups:
- All Treated Patients: All patients who were treated with protocol therapy
Arm/Group | All Treated Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of of Remission in Patients Who Receive GNKG168
Description: * MRD negative Complete Remission : Negative MRD (<0.01%), no evidence of circulating leukemic blasts or extramedullary disease, and recovery of peripheral counts (ANC ≥ 500/µL and PLT count ≥ 50,000 µL).
  * MRD negative Complete Remission without platelet recovery: Insufficient recovery of platelets (< 50,000/ µL) but otherwise meets the criteria of MRD-CR.
  * Stable Disease: Patient does not satisfy the criterion for PD, or has recovery of ANC ≥ 500/µL and fails to qualify for MRD-CR or MRD-CRp.
  * Progressive Disease: At least 5% of circulating leukemic cells or ≥5% in a marrow with count recovery, development of new sites of extramedullary disease, or other laboratory or clinical evidence of PD, with or without recovery of ANC or platelets.
  * Not evaluable: Patient does not satisfy the criterion for PD, and did not have a marrow evaluation, had inadequate marrow cell count, or had insufficient recovery of ANC for MRD-CR, MRD-CRp or SD classification.
Time Frame: Until patient is no longer being followed (off study)
Population: Study terminated early and the variable was not analyzed.
Arm/Group | All Treated Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the first dose of study therapy until 30 days after the last dose of study therapy. Therefore, for a given patient, AEs could be captured for 30-114 days depending on the length of time the patient received therapy.
Description: The definitions of AE and SAE do not differ from the clinicaltrials.gov definitions.
Groups:
- HSCT-Dose Level 0: Hematopoietic stem cell transplantation (HSCT)
  Dose level 0: 0.15 mg/kg/dose Dose level 1: 0.25 mg/kg/dose Dose level 2: 0.75 mg/kg/dose Dose level 3: 1.5 mg/kg/dose
- HSCT-Dose Level 1: Hematopoietic stem cell transplantation (HSCT)
  Dose level 1: 0.25 mg/kg/dose
- HSCT-Dose Level 2: Hematopoietic stem cell transplantation (HSCT)
  Dose level 2: 0.75 mg/kg/dose
- HSCT-Dose Level 3: Hematopoietic stem cell transplantation (HSCT)
  Dose level 3: 1.5 mg/kg/dose
- No HSCT-Dose Level 0: No Hematopoietic stem cell transplantation (HSCT)
  Dose level 0: 0.15 mg/kg/dose
- No HSCT-Dose Level 1: No Hematopoietic stem cell transplantation (HSCT)
  Dose level 1: 0.25 mg/kg/dose
- No HSCT-Dose Level 2: No Hematopoietic stem cell transplantation (HSCT)
  Dose level 2: 0.75 mg/kg/dose
- No HSCT-Dose Level 3: No Hematopoietic stem cell transplantation (HSCT)
  Dose level 3: 1.5 mg/kg/dose
Arm/Group | HSCT-Dose Level 0 | HSCT-Dose Level 1 | HSCT-Dose Level 2 | HSCT-Dose Level 3 | No HSCT-Dose Level 0 | No HSCT-Dose Level 1 | No HSCT-Dose Level 2 | No HSCT-Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0 | 0/0 | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0 | 0/0 | 1/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0 | 0/0 | 2/2 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSCT-Dose Level 0 (N=0) | HSCT-Dose Level 1 (N=1) | HSCT-Dose Level 2 (N=0) | HSCT-Dose Level 3 (N=0) | No HSCT-Dose Level 0 (N=0) | No HSCT-Dose Level 1 (N=2) | No HSCT-Dose Level 2 (N=0) | No HSCT-Dose Level 3 (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSCT-Dose Level 0 (N=0) | HSCT-Dose Level 1 (N=1) | HSCT-Dose Level 2 (N=0) | HSCT-Dose Level 3 (N=0) | No HSCT-Dose Level 0 (N=0) | No HSCT-Dose Level 1 (N=2) | No HSCT-Dose Level 2 (N=0) | No HSCT-Dose Level 3 (N=0)
Alanine aminotransferase increased (Investigations) | NA | NA | NA | NA | NA | 1 | NA | NA
Anemia (Blood and lymphatic system disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
Aspartate aminotransferase increased (Investigations) | NA | NA | NA | NA | NA | 1 | NA | NA
Creatinine increased (Investigations) | NA | NA | NA | NA | NA | 1 | NA | NA
Dyspepsia (Gastrointestinal disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
Edema limbs (General disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
Hypercalcemia (Investigations) | NA | NA | NA | NA | NA | 1 | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
Hyperkalemia (Investigations) | NA | NA | NA | NA | NA | 1 | NA | NA
Hypertension (Vascular disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
Hypokalemia (Investigations) | NA | NA | NA | NA | NA | 1 | NA | NA
Nausea (Gastrointestinal disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
Pain (General disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
Platelet count decreased (Investigations) | NA | NA | NA | NA | NA | 2 | NA | NA
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | NA | NA | NA | NA | NA | 1 | NA | NA
White blood cell decreased (Investigations) | NA | NA | NA | NA | NA | 1 | NA | NA

LIMITATIONS AND CAVEATS:
Early termination of study, due to SBI Biotech stopped supporting the study led to the small data set for analysis and technical problems with measurement leading to an uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days